CLINICAL TRIAL: NCT03563677
Title: Duale Lotsenstruktur Zur Abklärung Unklarer Diagnosen in Zentren für Seltene Erkrankungen
Brief Title: Dual Guidance Structure for Evaluation of Patients With Unclear Diagnosis in Centers for Rare Diseases
Acronym: ZSE-DUO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Hannover Medical School (Other); University Hospital, Aachen (Other); Allianz Chronischer Seltener Erkrankungen ACHSE e.V. (Unknown); Goethe University (Other); Universität Münster (Other); St. Josef Hospital Bochum (Other); Otto-von-Guericke University Magdeburg (Other); University Medical Center Mainz (Other); University Hospital Regensburg (Other); University Hospital Tuebingen (Other); University Hospital Ulm (Other); IKK gesund plus (Unknown); Techniker Krankenkasse (Other); University of Wuerzburg (Other); Universitätsklinikum Hamburg-Eppendorf (Other); AOK Hessen (Industry); LWL-Universitätsklinikum der Ruhr-Universität Bochum (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: ZSE-DUO_V1
Record Dates: First submitted 2018-05-23; First posted 2018-06-20 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Rare Diseases; Orphan Diseases
Keywords: psychosomatic; unclear diagnosis
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Intervention Model Description: Recruitment of 682 patients into control group during first 12 months of the project and, thereafter, recruitment of 682 patients during subsequent 12 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Standard evaluation process for patients approaching a center for rare diseases with an unclear diagnosis. The process includes the evaluation of complete medical records byan experienced physician, an outpatient visit to the center, and case discussion between experts. The process may also include an inpatient stay, a local case conference and a case conference between centers for rare diseases from different cities
- New Innovative Care (Experimental): The innovative evaluation process includes the additional involvement of a psychiatrists/psychosomatic expert in all of the processes described for the usual care arm plus the option to use telemedicine in the process of evaluation in addition to outpatient and inpatient visits and to transfer the patient back into standard care (i.e., primary care physician, rehabilitation, psychological/psychosomatic specialized care, etc.)
  Interventions: Other: dual expert guidance structure

INTERVENTIONS:
Other: dual expert guidance structure — Two medical experts, one somatic specialist and one psychiatrist/psychosomatic specialist see all medical records and the patients together
  Arms: New Innovative Care

SUMMARY:
In people suffering from a rare disease the diagnostic process and the confirmation of a final diagnosis is often ongoing for many years. Factors contributing to delayed diagnosis include the limited knowledge of health care professionals about rare diseases and their symptoms but also a psychiatric or psychosomatic (co-)morbidity obscuring the symptoms of the rare disease. The project ZSE-DUO will evaluate whether a combination of an expert in somatic medicine and a psychiatric/psychosomatic specialist will increase the rate of assured diagnoses in patients approaching a center of rare diseases (primary outcome), accelerate the process until a diagnosis is made, reduce the costs of diagnosing a patient, and lead to a higher satisfaction of patients and health care professionals. Furthermore, the project will evaluate whether the use of psychosomatic screening tools at registration of a patient in a center for rare diseases will help to guide the diagnostic process. Two cohorts of 682 patients each will be sequentially recruited over 9 plus 9 months: the Control group cohort (CG based on somatic expertise) and the Experimental group cohort (EG combined psychosomatic/somatic expertise Included will be persons from the age of at least 12 years presenting with symptoms and signs which are not explained by current diagnoses (as judged by the patient's primary care physician and a specialized physician at the center for rare diseases ZSE evaluating the medical records). Patients will be recruited from 11 German Centers for Rare Diseases associated with University hospitals in the cities of Aachen, Bochum, Frankfurt, Hannover, Magdeburg, Mainz, Münster, Regensburg, Tübingen, Ulm and Würzburg. Recruitment will be supported by a collaboration with the German patient organization representing many rare disease organizations ACHSE e.V. and a collaboration with the insurance companies Techniker Krankenkasse, IKK gesund plus and AOK Hessen who also provide data on costs of care. Data collection and analysis will be coordinated and performed by the Institute for Clinical Epidemiology and Biometry at the University of Würzburg, the Institute for Epidemiology, Social Medicine and Science of Health Care Systems in Hannover, and the Department of Medical Psychology in Hamburg. The project is funded by the Innovationsfond of the Federal Joint Committee in Germany.

ELIGIBILITY:
Inclusion Criteria:

* first contact with the Center for Rare Diseases for unclear diagnosis
* suspicion of a rare disease but no established diagnosis
* attending the Center for Rare Diseases as an outpatient
* written informed consent

Exclusion Criteria:

* age <12 years
* incomplete medical records including summary letters, imaging studies, blood tests etc.
* pre-diagnosed disease(s) explaining all symptoms

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1379 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Diagnoses made | 12 months after signing the consent form
  The number of diagnoses explaining the symptomatology of the patient made during the evaluation process

SECONDARY OUTCOMES:
Time to diagnosis | 12 months after signing the consent form
  The time it takes to make a diagnosis
Patient satisfaction with diagnostic process using ZUF-8 | 12 months after signing the consent form
  The patients' satisfaction with the diagnostic process is assessed in the total sample with the questionnaire ZUF-8 (Fragebogen zur Patientenzufriedenheit - patient satisfaction questionnaire) and in a randomly selected subsample of about 40 patients by structured telephone interviews.
Costs of the diagnostic process | up to 12 months after signing the consent from
  estimated costs from first contact with the center for rare diseases until a diagnosis explaining the symptoms has been established
Patients' quality of life using EQ-5D and SF12 (or KIDSCREEN-10 for children) | 12 months after signing the consent from
  Change in the patients' quality of life as assessed with the Quality of life questionnaires EQ-5D from the EuroQoL Group in all patients and Short Form 12 (SF-12) in patients 16 years and older. In patients younger than 16 years, the health-related quality of life questionnaire for children and adolescents KIDSCREEN-10 is used.
Physician satisfaction with new form of care using new questionnaire | 30 months after the project start (end of the intervention period)
  The satisfaction of physicians working in the Centers fro Rare Diseases with the new form of care compared to standard care will be assessed by a newly developed questionnaire administered to all physicians involved in patient care in the 11 centers. For the development of the questionnaire, 3 focus groups of 10 physicians each will be questioned.
Value of screening instruments for psychiatric-psychosomatic (co-)morbidities | 30 months after the project start (end of intervention period)
  Performance of screening tools to identify patients with psychiatric-psychosomatic comorbidities against the judgement of a psychiatrist/psychosomatic expert seeing the patient (intervention group only)

CONTACTS AND LOCATIONS:
Locations (12):
- Germany (12):
  - Center for Rare Diseases ZESE, University Hospital, Würzburg, Bavaria
  - Center for Rare Diseases ZSEA, University Hospital, Aachen
  - Center for Rare Diseases CeSER, St. Josef Hospital, Bochum
  - LWL-Universitätsklinikum der Ruhr-Universität, Bochum
  - Center for Rare Diseases FRZSE, UNiversity Hospital, Frankfurt
  - Center for Rare Diseases, Hannover Medical School, Hanover
  - Center for Rare Diseases MKSE, Otto von Guericke University, Magdeburg
  - Center for Rare Diseases, Medical Center, Mainz
  - Center for Rare Diseases, University Hospital, Münster
  - Center for Rare Diseases ZSER, University Hospital, Regensburg
  - Center for Rare Diseases, University Hospital, Tübingen
  - Center for Rare Diseases, University Hospital, Ulm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schippers C, Volk D, de Zwaan M, Deckert J, Dieris-Hirche J, Herpertz S, Schulz JB, Hebestreit H; ZSE-DUO Arbeitsgruppe. [ZSE-DUO - dual guidance structure at the centre for rare diseases]. Inn Med (Heidelb). 2022 Jul;63(7):791-797. doi: 10.1007/s00108-022-01350-8. Epub 2022 Jun 2. German. PMID 35925266
- [Background] Hebestreit H, Zeidler C, Schippers C, de Zwaan M, Deckert J, Heuschmann P, Krauth C, Bullinger M, Berger A, Berneburg M, Brandstetter L, Deibele A, Dieris-Hirche J, Graessner H, Gundel H, Herpertz S, Heuft G, Lapstich AM, Lucke T, Maisch T, Mundlos C, Petermann-Meyer A, Muller S, Ott S, Pfister L, Quitmann J, Romanos M, Rutsch F, Schaubert K, Schubert K, Schulz JB, Schweiger S, Tuscher O, Ungethum K, Wagner TOF, Haas K; ZSE-DUO working group. Dual guidance structure for evaluation of patients with unclear diagnosis in centers for rare diseases (ZSE-DUO): study protocol for a controlled multi-center cohort study. Orphanet J Rare Dis. 2022 Feb 14;17(1):47. doi: 10.1186/s13023-022-02176-1. PMID 35164804
- [Result] Hebestreit H, Lapstich AM, Brandstetter L, Krauth C, Deckert J, Haas K, Pfister L, Witt S, Schippers C, Dieris-Hirche J, Maisch T, Tuscher O, Barlescu L, Berger A, Berneburg M, Britz V, Deibele A, Graessner H, Gundel H, Heuft G, Lucke T, Mundlos C, Quitmann J, Rutsch F, Schubert K, Schulz JB, Schweiger S, Zeidler C, Zeltner L, de Zwaan M; ZSE-DUO Working Group. Effect of the addition of a mental health specialist for evaluation of undiagnosed patients in centres for rare diseases (ZSE-DUO): a prospective, controlled trial with a two-phase cohort design. EClinicalMedicine. 2023 Oct 6;65:102260. doi: 10.1016/j.eclinm.2023.102260. eCollection 2023 Nov. PMID 37855024
- [Result] Witt S, Kristensen K, Blomeke J, Hebestreit H, Wocker M, Pfister L, Bullinger M, Tuscher O, Deckert J, Graessner H, Lapstich AM, Zwaan M, Mundlos C, Quitmann JH. [Quality of Life and Experienced Distress of Patients Suspected of having a Rare (Chronic) Health Condition - Initial Findings from the ZSE-DUO Study]. Psychother Psychosom Med Psychol. 2023 Jan;73(1):9-15. doi: 10.1055/a-1814-3998. Epub 2022 Jul 6. German. PMID 35793670